CLINICAL TRIAL: NCT02130921
Title: Enhancing the Role of Commune Health Workers in HIV and Drug Control: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other)
Responsible Party: Principal Investigator, Li Li, PhD, Professor in Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA033609-01 (NIH)
Record Dates: First submitted 2014-05-01; First posted 2014-05-06 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Drug Dependence
Keywords: Stigma; HIV; CHWs; PLH; Injecting Drug Users; FM
MeSH Terms: conditions — Substance-Related Disorders; Social Stigma | interventions — Seroconversion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Community Health Workers (CHWs) in the control group will be invited to one group lecture didactically reviewing medical ethics, and the attending CHWs will be requested to pay a home visit to participating IDUs and FMs after the lecture.
- Intervention (Experimental): Intervention for CHWs: 3 sessions will cover the understanding stigma and its impact, self-protection and universal precaution adherence, effective communication with patients and family members, and motivational enhancement for behavioral change.
  Intervention for IDUs: CHWs who participate in the intervention will be required to conduct 3 individual sessions with participating IDUs covering the following topics: physical health, risk reduction behaviors, mental health, and community integration.
  Intervention for FMs: CHWs who participate in the intervention will be required to conduct 2 group sessions with participating FMs covering the following topics: healthy family routine, coping with caregiver burdens, enhance family relationships, support positive behavior change.
  Interventions: Behavioral: Intervention to Address Drug Use and HIV in Vietnam

INTERVENTIONS:
Behavioral: Intervention to Address Drug Use and HIV in Vietnam — Intervention for CHWs: 3 sessions will cover the understanding stigma and its impact, self-protection and universal precaution adherence, effective communication with patients and family members, and motivational enhancement for behavioral change.
  Intervention for IDUs: CHWs who participate in the intervention will be required to conduct 3 individual sessions with participating IDUs covering the following topics: physical health, risk reduction behaviors, mental health, and community integration.
  Intervention for FMs: CHWs who participate in the intervention will be required to conduct 2 group sessions with participating FMs covering the following topics: healthy family routine, coping with caregiver burdens, enhance family relationships, support positive behavior change.
  Arms: Intervention

SUMMARY:
This proposed study is an initiative for HIV prevention and care that integrates intervention efforts at multiple strata: Community Health Workers (CHWs), Injecting Drug Users (IDUs), and their Family Members (FMs). The proposed study will demonstrate the process of development, implementation, and evaluation of an intervention for CHWs, IDUs, and their FMs. One aim is to increase the CHWs' capacities to effectively interact with IDUs and FMs for HIV and drug use prevention and treatment. Using a combination of participatory action research and a randomized controlled trial design, this study has the potential to maximize PEPFAR impact in Vietnam and other PEPFAR-funded countries by identifying a sustainable mix of interventions and their implementation in different settings. The findings may benefit not only Vietnam but also a global audience by investigating enhanced methods for controlling the HIV epidemic.

DETAILED DESCRIPTION:
Vietnam is currently facing an HIV epidemic that had affected approximately 280,000 people by the end of 2009. Injecting Drug Use (IDU) is principal driver of the HIV epidemic, contributing to between 32 % and 58 % of all HIV cases in various provinces. However, it has proven difficult to address the needs of IDUs, a high-risk group, given the prevalence of stigmatization and drug use in Vietnamese society. In addition, Vietnamese people are highly family oriented and most young IDUs have daily family contact of live in their parents' homes. Thus the burden on the family is substantial, and even greater if the IDU is HIV+.

The study will be implemented in two provinces in Vietnam: Phu Tho and Vinh Phuc. A randomized controlled trial will be conducted to evaluate the impact of the intervention in 60 commune health centers. From each center we will recruit 5 Community Health Workers (CHWs), 15 Injecting Drug Users (IDUs), and 10 Family Members (FMs) (totaling 300 CHWs, 900 IDUs, and 600 FMs). The outcomes will be evaluated at 3-, 6-, 9-, and 12- month follow-up assessments. The specific aims of the study are as follows:

1. To develop and implement an integrated intervention, CHW CARE, for CHWs, IDUs, and their FMS in Vietnam
2. To evaluate the feasibility and operational procedures of the intervention with an implementation pilot, including process evalution and monitoring, and participants feedback.
3. To assess the impact of the intervention by comparing outcome measures of CHWs, IDUs, and FMs in the intervention group to those in the control group.
4. To explore the relationships between the intervention outcomes of CHWs, IDUs, and FMs.

ELIGIBILITY:
Inclusion Criteria:

Injecting Drug Users:

* Age 18 or over
* Having a history of drug use
* Currently residing in the selected commune, and have no plan to move to other communes in the following year
* Voluntary informed consent

Family members of Injecting Drug Users:

* Age 18 or over
* Immediate or extended family member of the Injecting Drug User.
* Previous knowledge of the drug use of the IDU.
* Voluntary informed consent
* Currently residing in the selected commune, and have no plan to move to other communes in the following year

Community Health Workers:

* Age 18 or over
* Doctor, nurse, or other care provider working at the selected commune health centers
* Informed consent

Exclusion Criteria:

Injecting Drug Users:

* Those who have psychosis or neurological damage, or cannot understand the study purposes as judged by the interviewer in consultation with a clinic supervisor, will be excluded
* Does not meet other inclusion criteria

Family members of Injecting Drug Users:

* Those who have psychosis or neurological damage, or cannot understand the study purposes as judged by the interviewer in consultation with a clinic supervisor, will be excluded
* Does not meet other inclusion criteria

Community Health Workers:

* Inability to give informed consent
* Does not meet other inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Community Health Worker (CHW) Interaction with patients | Changes from baseline to 3-, 6-, 9- and 12- month follow-up
  Provider-Client interaction scale will be used.
Injecting Drug User (IDU) drug use | baseline, 3-, 6-, 9- and 12- month follow-up
  Urine test results

SECONDARY OUTCOMES:
Community Health Worker (CHW) job safety, support, and satisfaction | Changes from baseline to 3-, 6-, 9-, and 12- month follow-up
  This will be assessed by perceived risk at work and institutional support. Additionally by job satisfaction using a 29-item scale.
Community Health Worker (CHW) knowledge and adherence to universal precautions | Changes from baseline to 3-, 6-, 9-, and 12- month follow-up
  This will be assessed with the universal precautions knowledge scale.
Injecting Drug User (IDU) family and social support | Changes from baseline to 3-, 6-, 9- and 12- month follow-up
  This is measured by two instruments. Social Support Questionnaire (Short; SSQ6) is a 6-item assessment to measure satisfaction of social support. Number of social support providers is captured up to 9 people in various support dimensions (Sarason et al., 1983). Medical Outcomes Study- Social Support Scale (MOS-SS) is a 20-item scale that measures the strength of perceived social support available. The scale consists of five dimensions: emotional support, informational support, tangible support, positive social interaction, and affection
Family Member (FM) social support | Changes from baseline to 3-, 6-, 9-, and 12- month follow-up
  This is measured by two instruments. Social Support Questionnaire (Short; SSQ6) is a 6-item assessment to measure satisfaction of social support. Number of social support providers is captured up to 9 people in various support dimensions (Sarason et al., 1983). Medical Outcomes Study- Social Support Scale (MOS-SS) is a 20-item scale that measures the strength of perceived social support available. The scale consists of five dimensions: emotional support, informational support, tangible support, positive social interaction, and affection.
Community Health Worker (CHW) general prejudicial attitude | Changes from baseline to 3-, 6-, 9- and 12- month follow-up
  A scale will be used
Family Member (FM) Caregiver burden/coping | Changes from baseline to 3-,6-,9-, and 12-month follow-up
  Caregiver burden and coping scales will be used

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, Ph.D, Principal Investigator — University of California, Los Angeles
Locations (2):
- Vietnam (2):
  - Phú Thọ commune health centers, Phú Thọ
  - Vĩnh Phúc commune health centers, Vĩnh Phúc